## Testing Effectiveness of a Peer-Led Intervention to Enhance Community Integration

NCT02508480

Statistical Analysis Plan

Date: July 24th, 2019

## Statistical Analysis Plan-

Intent-to-treat analyses will be conducted on the full sample of participants, regardless of actual exposure to the Photovoice program. Based on our pilot RCT study of Photovoice we are confident that majority of participants randomized to the Photovoice group will receive the intervention. However, if significant rates of non-exposure occur, we will also conduct separate analyses on treatment exposed participants. The intent-to-treat sample will include all participants for whom we have baseline data. It assumes that participants who are not exposed to the Photovoice program are not also study dropouts, and thus the analyses will include all available study participants. These analyses are the primary gauge of the effectiveness of the Photovoice program. If dropout rates from the Photovoice group exceed 20% we will explore the question of treatment effectiveness for those who participated in the Photovoice program. Participants will be classified based on their level of participation, with "exposure" defined as attendance at more than one-half of the 10 sessions (6 or more), with parallel analyses comparing the exposed Photovoice group with SAU. We will test the following primary hypotheses:

Hypothesis 1: Compared to SAU, clients randomized to the Photovoice program will demonstrate significantly greater improvements at post-treatment and 3- and 6-month follow-ups in their capacity to resist public prejudice and discrimination, including reduced self-stigma and perceived stigma, and increased proactive coping with public prejudice and discrimination (e.g., confronting prejudicial and discriminatory attitudes and behaviors). We will test this hypothesis by using the total score on the Internalized Stigma of Mental Illness Scale<sup>78</sup> and on the Stigma Scale<sup>93</sup>, and the sum of the two proactive coping subscales on the Coping with Stigma Scale (Educating Others, Challenging Others)<sup>92</sup> and fitting covariance pattern models (using SAS PROC MIXED) and examining time (baseline, post-treatment, 3- and 6 month follow-ups), group, and the group by time interaction effects.

Hypothesis 2: Compared to SAU, clients randomized to Photovoice will show significantly greater improvements at post-treatment and 3- and 6- month follow-ups in community functioning and integration. The scores on the Temple University Community Participation Scale will be used as measures of community integration.